CLINICAL TRIAL: NCT03917017
Title: The Evaluation of Surgical Decisions and Prognosis of the Radiomics and Watson Artificial Intelligence in Patients With Hepatocellular Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201901
Record Dates: First submitted 2019-04-04; First posted 2019-04-16 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Liver Resection
Keywords: radiomics; Watson artificial intelligence; hepatocellular carcinoma; surgical decisions; prognosis
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Radiomics

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radiomics and Watson artificial intelligence (Experimental)
  Interventions: Device: Radiomics and Watson artificial intelligence

INTERVENTIONS:
Device: Radiomics and Watson artificial intelligence — The artificial intelligence platform developed by IBM Watson can provide treatment decisions and corresponding theoretical basis to guide surgical decisions based on the key clinical data of liver cancer patients.
  The imaging histology can be used to conduct intraoperative navigation surgical resection and treatment monitoring, and established a prognosis model to predict the prognosis of patients by grading the results of postoperative follow-up and microvascular invasion of pathological liver cancer, so as to better achieve accurate diagnosis and treatment of the disease.

SUMMARY:
The aim of this study was to evaluate the surgical decisions and prognosis of the radiomics and Watson artificial intelligence in patients with hepatocellular carcinoma.

DETAILED DESCRIPTION:
Hepatectomy is an effective treatment for patients with hepatocellular carcinoma, but liver failure after hepatectomy may lead to increased postoperative mortality.Therefore, it is very important to make preoperative surgical decisions, evaluate the safety of the operation and identify which patients are likely to suffer from liver failure.Imaging omics is a newly emerging research method in recent years, which has great potential in cancer diagnosis and treatment, and can monitor treatment and predict the prognosis of patients, so as to better realize accurate diagnosis and treatment of diseases.The artificial intelligence platform developed by IBM Watson for Watson tumor treatment decisions can provide treatment decisions and corresponding theoretical basis to guide surgical decisions based on the key clinical data of liver cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years≤ Age ≤80 years
2. Compling with the diagnosis criteria of complex hepatic carcinoma.
3. Primary hepatic carcinoma without intrahepatic or extrahepatic extensive cancer metastasis, the metastatic hepatic carcinoma whose primary focal has been controlled
4. Preoperative liver function is Child - Pugh grade A or B.
5. The patients are volunteered for the study.

Exclusion Criteria:

1. Patients with mental illness.
2. Patients can't tolerate the operation owe to a variety of basic diseases (such as severe cardiopulmonary insufficiency, renal insufficiency, cachexia and blood system diseases, etc.)
3. The patients refused to take part in the study.
4. There are other co-existed malignant tumors.
5. Benign liver diseases.
6. Indocyanine green allergy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative survival | 5 years
  Survival after hepatectomy

SECONDARY OUTCOMES:
Disease-free survival | 5 years
  Survival time without tumor after HCC resection

OTHER OUTCOMES:
Intraoperative blood loss | intraoperative
  Operative outcome

CONTACTS AND LOCATIONS:
Overall Officials: Chihua Fang, M.D;Ph.D, Study Director — China, Guangdong Zhujiang Hospital of The Southern Medical University
Locations (1):
- Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong, China